CLINICAL TRIAL: NCT06754449
Title: The Effect of Painting Therapy on Visual Perception, Hand Functions, Social Participation and Quality of Life in Children
Brief Title: The Effect of Painting Therapy in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Nilay Şahan, Principle Investigator, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ae2036af3d594ea0
Record Dates: First submitted 2024-12-13; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Child Development; Art Therapy
Keywords: art therapy; visual perception; hand skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The children in the control group should not have participated in any painting course.
- Art therapy group (Experimental): The children in the art therapy group will receive painting and drawing-based painting therapy for 4 weeks, 2 days a week for 1 hour.
  Interventions: Other: Art therapy group

INTERVENTIONS:
Other: Art therapy group — Application of different applications of art therapy such as painting, drawing, cutting to children
  Arms: Art therapy group

SUMMARY:
This study was designed to examine the effect of picture supported art therapy on visual perception, hand functions, participation and quality of life of children in healthy children.

DETAILED DESCRIPTION:
It is planned that at least 25 children in each group will participate in the study. For both the control group and the study group, the sample of the study will consist of children between the ages of 6-12 who do not have any known disease/disability and show typical development, who voluntarily agree to participate in our study and sign the consent form. In addition, children in the control group should not have participated in any art course.Sociodemographic information will be asked first in the evaluation of the individuals in the study. Then, which hand of the children is dominant will be determined with Edinburg Hand Preference Questionnaire. Visual perception of the children will be evaluated with the shape-ground subtest of the Ayres Southern California Sensory Integrity Test, hand skills will be evaluated with the 9-hole peg test and the sense of kinesthesia in their fingers will be evaluated with the kinesthesia subtest of the Ayres Southern California Sensory Integrity Test. Children's quality of life will be assessed with the Young Child Quality of Life Questionnaire in accordance with their age. The Child and Adolescent Participation Questionnaire will be given to the parents to question the social participation of the children and the Conners Parent Rating Scale will be given to the parents to evaluate the disruptive behaviour disorders. Initial assessments will be made both in the study group and in the control group.The children in the study group will receive painting and drawing-based art therapy for 4 weeks, 2 days a week for 1 hour. After 4 weeks, all evaluations will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* The sample of the study for both the control group and the study group,
* To be between 6-12 years old,
* not having any known illness/disability
* voluntarily agree to participate in our study
* The children in the control group should not have participated in any art course.

Exclusion Criteria:

* The sample of the study for both the control group and the study group,
* Not to be between 6-12 years old
* having any known illness/disability (such as neurological, mental illness)
* not voluntarily agreeing to participate in our study
* Children in the control group participated in any art course

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Children's age | Day 1 of the study will be evaluated.
  age in year

SECONDARY OUTCOMES:
Children's weight | Day 1 of the study will be evaluated.
  weight in kilograms
Children's height | Day 1 of the study will be evaluated.
  height in meters
Childern's body mass index (BMI) | Day 1 of the study will be evaluated.
  weight and height will be combined to report BMI in kg/m2
Mothers' age | Day 1 of the study will be evaluated.
  age in year
Mothers' education status | Day 1 of the study will be evaluated.
  education status like primary school, high school, university, etc.
visual perception | From enrollment to the end of treatment at 4 weeks.
  Children's visual perception will be assessed using the shape-ground subtest of the Ayres Southern California Sensory Integrity Test. Ayres Southern California Sensory Integrity Tests is a standardised and reliable test battery consisting of 17 subtests and can be used in both children and adults from the age of 4.
Hand function | From enrollment to the end of treatment at 4 weeks.
  Individuals' manual dexterity will be assessed with the 9-Hole Peg Test. It is a quick simple manual dexterity test that is particularly sensitive to changes in upper extremity performance. The test material consists of 9 small sticks made in standard sizes and a board with 9 holes on which they are placed. Individuals are asked to place the sticks one by one on the board as fast as possible and then remove them. Time is measured with a stopwatch. Measurement is performed for both extremities, first the right and then the left hand.
Hand preference | From enrollment to the end of treatment at 4 weeks.
  It is a frequently applied questionnaire to determine the dominant hand. It questions the hand or hands used in 10 activities of daily living such as writing, drawing, throwing, using scissors, using a toothbrush, using a knife without a fork, using a spoon, sweeping with a broom, lighting a match and opening a box. The scoring ranges from -100 (left hand) to +100 (right hand). The evaluation is calculated with the Geschwind Score (GS). In the scoring; those with a score of 80 to 100 are defined as strong right-handed, those with a score of 20 to 75 as weak right-handed, those with a score of -15 to 15 as mixed-handed, those with a score of -20 to -75 as weak left-handed and those with a score of -80 to -100 as strong left-handed.
kinesthesia assessment | From enrollment to the end of treatment at 4 weeks.
  Ayres Southern California Sensory Integrity Tests is a standardized and reliable test battery consisting of 17 subtests and can be used in both children and adults from the age of 4 years. It was developed by Anne Jean Ayres in 1979 to examine sensory processing skills for different conditions such as vestibular, proprioceptive, kinesthetic and tactile systems and to reveal inadequate function in the sensory processing process. In our study, the kinesthesia subtest of the Ayres Southern California Sensory Integrity Tests will be used.
The Child and Adolescent Participation Questionnaire | From enrollment to the end of treatment at 4 weeks.
  The Child and Adolescent Participation Questionnaire is a questionnaire used to assess social participation. The CASP scale assesses the child's participation in the home, school, neighborhood and community. It consists of a total of 20 questions and has 4 sub-sections. Home participation consists of 4 questions, school participation consists of 5 questions, neighborhood and community participation consists of 4 questions, and home and community activities consists of 5 questions. The participation questionnaire is completed by the child's family or carers. The evaluation is based on a total of 100 points. Low scores indicate a low level of participation; high scores indicate a good level of participation. Scoring is done between 0-4.
Young Child Quality of Life Questionnaire | From enrollment to the end of treatment at 4 weeks.
  The scale aims to measure the general quality of life in the 2-18 age group. The scale consists of a total of 23 questions including physical function 8 questions, emotional function 5 questions, social function 5 questions and school function 5 questions and was prepared for four different age groups.Firstly, the total scale score (TTS), secondly, the total physical health score (FSTP), and thirdly, the total psychosocial health score (PSTP), which consists of the calculation of item scores evaluating emotional, social and school functionality, are calculated. The items are scored between 0-100.The higher the total score of the scale, the better the health-related quality of life is perceived.
Revised Conners Parent Rating Scale Short Turkish Form | From enrollment to the end of treatment at 4 weeks.
  It is a scale used to screen 'Attention Deficit and Disruptive Behavior Disorders'. High scores obtained from the scale indicate the intensity of symptoms specific to destructive disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Şahan, PhD, Study Director — Çankırı Karatekin University

IPD SHARING:
Plan to Share IPD: Yes
The data that support the ﬁndings of this study will be available upon reasonable request but will not be publicly accessible due to privacy or conﬁdentiality concerns.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately following publication.No end date.
Access Criteria: Proposals should be directed to nilaysahan@karatekin.edu.tr.